CLINICAL TRIAL: NCT05046457
Title: Beta-Cryptoxanthin (BCX) Supplementation and Circulating Carotenoid Concentrations in Women: A Randomized, Controlled, Double-blinded and 8 Week Parallel Trial
Brief Title: Beta-cryptoxanthin Supplement: Absorption and Function
Acronym: BETA+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Human Development and Potential (IHDP), Singapore (Other)
Collaborators: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Principal Investigator, Karen Tan Mei Ling, Research Clinician, Institute for Human Development and Potential (IHDP), Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2021/00455
Record Dates: First submitted 2021-08-23; First posted 2021-09-16 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Beta-cryptoxanthin Supplementation
Keywords: Beta-cryptoxanthin; Supplementation; Carotenoids; Bioavailability
MeSH Terms: interventions — Beta-Cryptoxanthin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 3mg BCX supplement (Experimental): One 3mg BCX capsule + one placebo capsule to be taken once per day for 8 weeks
  Interventions: Dietary Supplement: Beta-cryptoxanthin (BCX)
- 6mg BCX supplement (Experimental): Two 3mg BCX capsules to be taken once per day for 8 weeks
  Interventions: Dietary Supplement: Beta-cryptoxanthin (BCX)
- 0mg BCX supplementation (Placebo Comparator): Two placebo capsules to be taken once per day for 8 weeks
  Interventions: Dietary Supplement: Beta-cryptoxanthin (BCX)

INTERVENTIONS:
Dietary Supplement: Beta-cryptoxanthin (BCX) — Subjects will be randomised into one of the three study treatment arms.

SUMMARY:
Beta-cryptoxanthin (BCX) is a naturally occurring member of the carotenoid family, found in a wide range of fruits and vegetables. The unique biological functions of BCX have not been well-established, although BCX, like other members of the carotenoids have antioxidant functions. BCX, may also serve as a precursor of Vitamin A. Vitamin A has a wide range of functions including maintain immunity, vision, growth and development. Whilst not specific for BCX, epidemiological studies indicate that dietary intake of carotenoids may be of benefit in maintaining cognitive health and reducing stress via its antioxidant, anti-inflammatory and immunomodulatory properties. This pilot study aims to establish the relationship between supplemental dose and circulating concentrations of BCX and related carotenoids in circulation. Results obtained from this study will provide greater insight of bioavailability and carotenoid metabolism, necessary for larger supplementation in selected target populations.

DETAILED DESCRIPTION:
In previous Singapore maternal and child health cohort study, Growing up towards healthy outcomes (GUSTO), it established potentially significant health function to be significantly correlated with BCX. At childbirth, mothers' blood concentrations of carotenoids, including α-, β-carotene and BCX were simultaneously measured by ultra-performance liquid chromatography. Unique to the carotenoids, there was a correlation between higher maternal plasma concentrations of BCX with lower rates of depression and reduced anxiety scores during pregnancy for the mother. Furthermore, the concentrations of BCX were uniquely correlated with child neurocognitive function by age 2 years.

Current studies have only been food-based efficacy trials with an increase of dietary BCX intake through BCX-rich foods in humans. There have been no direct assessments of risk associated with BCX exposure, and current evidence in the literature does not identify any consistent, substantial risks for any level of BCX supplementation. Overall, the utility of BCX as a pro-vitamin A is clear, but evidence towards benefits beyond this role is inconsistent.

Hence, this is a pilot study that will aim to examine bioavailability of a novel BCX preparation supplemented at 2 doses (3mg and 6mg daily) versus placebo, consumed once daily in a randomised, doubled-blinded parallel trial, in healthy female subjects of reproductive age.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 21 - 35 years old, residing in Singapore
2. Body mass index (BMI) between 18.5 to 27.5 kg/m2
3. Subject should not be pregnant or breastfeeding during study period
4. Subject should not be planning to conceive within 3 months from enrolment
5. Subject must voluntarily consent to participate in this study and provide their written informed consent prior to start of study
6. Subject is always willing to comply with study regulations and instructions

Exclusion Criteria:

1. Any current diagnosis or history of cardiovascular, hepatic, renal, metabolic (e.g. diabetes), immunological, gastrointestinal diseases, psychiatric disorders or chronic diseases
2. Participation in another simultaneous clinical study
3. Ongoing adherence to weight reduction diet and/or programs
4. Use of medication and supplementation with other carotenoids reasonable expected to impact on primary outcome (e.g. drug treatment for hyperlipidemia)
5. A history of drug abuse
6. Current smoker or excessive alcohol intake (>4 standard drinks per day)
7. Subject has a known allergy or sensitivity to BCX or any ingredients of the study products provided

Ages: 21 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in plasma concentration of BCX over 8 weeks | Baseline, Week 2, Week 4, Week 8
  Fasting plasma carotenoids concentrations

SECONDARY OUTCOMES:
Height measurement | Baseline
  Height in centimeters (cm)
Change in weight | Baseline, Week 8
  Weight in kilograms (kg)
Change in Body Mass Index (BMI) | Baseline, Week 8
  BMI in kg/m^2 (from converted height in centimeters to meters)
Change in waist circumference | Baseline, Week 8
  Waist circumference in centimeters (cm)
Change in body composition - Total body fat | Baseline, Week 8
  Body fat analysis in percentage (%)
Changes in General Health Questionnaire (GHQ-12) scores | Baseline, Week 8
  - GHQ-12 scores for measure of physiological distress
Change in Pittsburgh Sleep Quality Index (PSQI) scores | Baseline, Week 8
  - PSQI scores for measures of sleep quality and patterns
Change in State-Trait Anxiety Inventory (STAI) scores | Baseline, Week 8
  - STAI scores for measures of anxiety
Change in Perceived Stress Scale (PSS) scores | Baseline, Week 8
  - PSS scores for measures of stress perceptions
Change in Quality of Life Enjoyment and Satisfaction Questionnaire (QLES) scores | Baseline, Week 8
  - QLES scores for measures of the degree of life satisfaction
Change in Satisfaction with Life Scale (SLS) scores | Baseline, Week 8
  - SLS scores for measures of subjective well-being
Change in Depression Anxiety Stress Scales (DASS) scores | Baseline, Week 2, Week 4, Week 8
  - DASS scores for measures of the negative emotional states of depression, anxiety and stress
Change in gut microbiota composition | Baseline, Week 8
  - Assessed by 16S rRNA gene sequencing of stool sample
Change in sleep/wake time | Baseline, Week 8
  - Assessed with 7 consecutive days of total sleep time and wake after sleep onset measured using a wrist worn accelerometer
Change in physical activity | Baseline, Week 8
  - Assessed with 7 consecutive days of raw acceleration, steps taken and activity counts measured using a wrist worn accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tan Mei Ling, PhD, Principal Investigator — Institute for Human Development and Potential (IHDP), Singapore
Locations (1):
- Singapore Institute for Clinical Sciences, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No